CLINICAL TRIAL: NCT06918730
Title: Prospective Randomized Controlled Trial (RCT)Comparing Clinical Outcomes Between Underwater Versus Carbon Dioxide Insufflation During Peroral Endoscopic Myotomy (U-POEM Trial)
Brief Title: U-POEM vs CO2-POEM
Acronym: U-POEM
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: AdventHealth (Other)
Collaborators: Mayo Clinic (Other); University of South Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2263975
Record Dates: First submitted 2025-03-21; First posted 2025-04-09 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2025-03

CONDITIONS: Esophageal Motility Disorders
Keywords: POEM; U-POEM; CO2-POEM; Esophageal motility
MeSH Terms: conditions — Esophageal Motility Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CO2-POEM (Experimental): POEM is routinely performed under carbon dioxide insufflation (CO2-POEM) as this gas is more rapidly absorbed than air.
  Interventions: Procedure: CO2-POEM
- U-POEM (Experimental): Water immersion for luminal distension of the GI tract as opposed to carbon dioxide insufflation
  Interventions: Procedure: U-POEM

INTERVENTIONS:
Procedure: U-POEM — Water immersion for luminal distension of the GI tract as opposed to carbon dioxide insufflation
  Arms: U-POEM
Procedure: CO2-POEM — POEM is routinely performed under carbon dioxide insufflation (CO2-POEM) as this gas is more rapidly absorbed than air.
  Arms: CO2-POEM

SUMMARY:
Multicenter randomized trial comparing post-procedural pain intensity after Per-Oral endoscopic myotomy (POEM) between two types of standard of care insufflation methods (CO2 vs Underwater).

POEM is routinely performed under carbon dioxide insufflation (CO2-POEM) as this gas is more rapidly absorbed than air, which has been shown to reduce gas-related complications.

Water immersion for luminal distension of the GI tract as opposed to carbon dioxide insufflation has been shown to be associated with improved patient satisfaction, safety profile and even higher detection of polyps during colonoscopy in randomized trials

Aim 1. The primary aim is to compare post-procedural pain following U-POEM vs. CO2-POEM.

Aim 2. Compare the proportion of patients that require post-procedural admission for pain management.

Aim 3. Compare the need for analgesic medications for pain control in patients undergoing U-POEM vs. CO2-POEM.

Aim 4. Compare technical and clinical success between U-POEM vs. CO2-POEM. Technical success is defined as successful completion of the procedure whereas clinical success will be defined as an Eckardt score ≤ 3 at the time of follow-up.

Aim 5. Compare and evaluate procedural characteristics between the two groups.

1. Compare procedural time between U-POEM and CO2-POEM.
2. Compare the mean number of coagulations with hemostatic forceps for active intraprocedural bleeding and the mean number of times in which a device besides an electrosurgical knife was required for prophylactic ablation of vessels.
3. Adverse event rate (i.e. bleeding, perforation).

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Ability to provide informed consent
* Patient scheduled to undergo POEM procedure for esophageal dysmotility

Exclusion Criteria:

* Inability to provide informed consent
* Any contraindication to POEM as per the endoscopist at the time of endoscopic evaluation (example: esophageal stricture, malignancy).
* Any standard contraindication, including pregnancy, to anesthesia and/or colonoscopy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2025-05-23 (Actual); Primary Completion 2025-10-30 (Actual); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Pain measurement outcomes post procedure: Numeric Pain Scale | Through study completion. Before Endoscopic Procedure (Day 1), Post Endoscopic Procedure (Day 1), and follow-up visit (Up to 6 months post procedure)
  The primary aim is to compare post-procedural pain following U-POEM vs. CO2-POEM.
  Using Numeric Pain Scale (NPS)
  NPS is a numeric scale ranging from 0 (no pain) to 10 (worst pain imaginable)
Pain measurement outcomes post procedure: Pain Quality Assessment Scale | Through study completion. Before Endoscopic Procedure (Day 1), Post Endoscopic Procedure (Day 1), and follow-up visit (Up to 6 months post procedure)
  The primary aim is to compare post-procedural pain following U-POEM vs. CO2-POEM.
  Pain Quality Assessment Scale (PQAS).
  PQAS is a numeric scale ranging from 0 (no pain) to 10 (worst pain imaginable)

SECONDARY OUTCOMES:
Readmission rate | 30 days post procedure (+- 7 days)
  Compare the proportion of patients that require post-procedural admission for pain management.
Analgesic medication needs | 30 days post procedure (+- 7 days)
  Compare the need for analgesic medications for pain control in patients undergoing U-POEM vs. CO2-POEM through electronic medical records.
Compare technical success between POEM procedures | up to 6 months
  Compare clinical success between U-POEM vs. CO2-POEM. Clinical success will be defined as an Eckardt score ≤ 3 at the time of follow-up.
  Achalasia Severity is measured by the Eckardt Score which consists of 4 questions used to characterize the severity of achalasia.
  The questions include symptoms related to:
  * Dysphagia
  * Chest pain
  * Regurgitation
  * Weight loss.
  Each question is assigned a score from 0 to 3 based on the patient's self-reported response.
  The overall score ranges from 0-12, with anything less than 3 meaning no active symptoms, and anything higher than a 3 suggestive of active symptoms.
Compare technical success between POEM procedures | up to 6 months
  Compare technical success between U-POEM vs. CO2-POEM. Technical success is defined as successful completion of the procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Dennis Yang, MD, Principal Investigator — AdventHealth Medical Group
Locations (1):
- AdventHealth Orlando, Orlando, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ponds FA, Fockens P, Lei A, Neuhaus H, Beyna T, Kandler J, Frieling T, Chiu PWY, Wu JCY, Wong VWY, Costamagna G, Familiari P, Kahrilas PJ, Pandolfino JE, Smout AJPM, Bredenoord AJ. Effect of Peroral Endoscopic Myotomy vs Pneumatic Dilation on Symptom Severity and Treatment Outcomes Among Treatment-Naive Patients With Achalasia: A Randomized Clinical Trial. JAMA. 2019 Jul 9;322(2):134-144. doi: 10.1001/jama.2019.8859. PMID 31287522
- [Background] Werner YB, Hakanson B, Martinek J, Repici A, von Rahden BHA, Bredenoord AJ, Bisschops R, Messmann H, Vollberg MC, Noder T, Kersten JF, Mann O, Izbicki J, Pazdro A, Fumagalli U, Rosati R, Germer CT, Schijven MP, Emmermann A, von Renteln D, Fockens P, Boeckxstaens G, Rosch T. Endoscopic or Surgical Myotomy in Patients with Idiopathic Achalasia. N Engl J Med. 2019 Dec 5;381(23):2219-2229. doi: 10.1056/NEJMoa1905380. PMID 31800987
- [Background] Yang D, Bechara R, Dunst CM, Konda VJA. AGA Clinical Practice Update on Advances in Per-Oral Endoscopic Myotomy (POEM) and Remaining Questions-What We Have Learned in the Past Decade: Expert Review. Gastroenterology. 2024 Dec;167(7):1483-1490. doi: 10.1053/j.gastro.2024.08.038. Epub 2024 Oct 16. PMID 39425737
- [Background] Reddy CA, Tavakkoli A, Abdul-Hussein M, Almazan E, Vosoughi K, Ichkhanian Y, Al-Hawary M, Chang AC, Chen JW, Korsnes S, Elmunzer BJ, Khashab MA, Law R. Clinical impact of routine esophagram after peroral endoscopic myotomy. Gastrointest Endosc. 2021 Jan;93(1):102-106. doi: 10.1016/j.gie.2020.05.046. Epub 2020 Jun 3. PMID 32504702
- [Background] Benias PC, Korrapati P, Raphael KL, D'Souza LS, Inamdar S, Trindade AJ, Lee C, Kumbhari V, Sejpal DV, Okolo P, Khashab MA, Miller L, Carr-Locke D. Safety and feasibility of performing peroral endoscopic myotomy as an outpatient procedure with same-day discharge. Gastrointest Endosc. 2019 Oct;90(4):570-578. doi: 10.1016/j.gie.2019.04.247. Epub 2019 May 10. PMID 31078571
- [Background] Cloutier Z, Mann A, Doumouras AG, Hong D. Same-day discharge is safe and feasible following POEM surgery for esophageal motility disorders. Surg Endosc. 2021 Jul;35(7):3398-3404. doi: 10.1007/s00464-020-07781-4. Epub 2020 Jul 9. PMID 32648037
- [Background] Maeda Y, Hirasawa D, Fujita N, Obana T, Sugawara T, Ohira T, Harada Y, Yamagata T, Suzuki K, Koike Y, Yamamoto Y, Kusaka Z, Noda Y. A pilot study to assess mediastinal emphysema after esophageal endoscopic submucosal dissection with carbon dioxide insufflation. Endoscopy. 2012 Jun;44(6):565-71. doi: 10.1055/s-0031-1291664. Epub 2012 Mar 9. PMID 22407383
- [Background] Pannu D, Yang D, Abbitt PL, Draganov PV. Prospective evaluation of CT esophagram findings after peroral endoscopic myotomy. Gastrointest Endosc. 2016 Sep;84(3):408-15. doi: 10.1016/j.gie.2016.02.022. Epub 2016 Feb 22. PMID 26907745
- [Background] Lee JY, Lim CH, Kim DH, Jung HY, Youn YH, Jung DH, Park JC, Moon HS, Hong SJ; Therapeutic Endoscopy and Instrument for Functional Gastrointestinal Disorders Study Group Under the Korean Society of Neurogastroenterology and Motility. Adverse Events Associated With Peroral Endoscopic Myotomy Affecting Extended Hospital Stay: A Multi-center Retrospective Study in South Korea. J Neurogastroenterol Motil. 2022 Apr 30;28(2):247-254. doi: 10.5056/jnm21081. PMID 35362451
- [Background] Cadoni S, Gallittu P, Sanna S, Fanari V, Porcedda ML, Erriu M, Leung FW. A two-center randomized controlled trial of water-aided colonoscopy versus air insufflation colonoscopy. Endoscopy. 2014 Mar;46(3):212-8. doi: 10.1055/s-0033-1353604. Epub 2013 Nov 11. PMID 24218307
- [Background] Hsieh YH, Koo M, Leung FW. A patient-blinded randomized, controlled trial comparing air insufflation, water immersion, and water exchange during minimally sedated colonoscopy. Am J Gastroenterol. 2014 Sep;109(9):1390-400. doi: 10.1038/ajg.2014.126. Epub 2014 Jun 3. PMID 24890443
- [Background] Binmoeller KF, Bhat YM. Underwater peroral endoscopic myotomy. Gastrointest Endosc. 2016 Feb;83(2):454. doi: 10.1016/j.gie.2015.08.066. Epub 2015 Sep 8. No abstract available. PMID 26358328
- [Background] Uchima H, Colan J, Marin I, Moreno V, Larios G, Tazi R, Serra J. Underwater peroral endoscopic myotomy (u-POEM) after tension capnoperitoneum and capnothorax during POEM. Endoscopy. 2020 Nov;52(11):E396-E397. doi: 10.1055/a-1144-2547. Epub 2020 Apr 17. No abstract available. PMID 32303086
- [Background] Capogreco A, de Sire R, Massimi D, Alfarone L, Maselli R, Hassan C, Repici A. Underwater coagulation using hybrid knife in peroral endoscopic myotomy for achalasia. Endoscopy. 2024 Jul;56(7):547-548. doi: 10.1055/a-2292-8460. Epub 2024 Jun 27. No abstract available. PMID 38936349
- [Background] Yang D, Pannu D, Zhang Q, White JD, Draganov PV. Evaluation of anesthesia management, feasibility and efficacy of peroral endoscopic myotomy (POEM) for achalasia performed in the endoscopy unit. Endosc Int Open. 2015 Aug;3(4):E289-95. doi: 10.1055/s-0034-1391965. Epub 2015 May 5. PMID 26357672
- [Background] Sarkar S, Khanna P, Gunjan D. Anesthesia for Per-oral endoscopic myotomy (POEM) - not so poetic! J Anaesthesiol Clin Pharmacol. 2022 Jan-Mar;38(1):28-34. doi: 10.4103/joacp.JOACP_179_20. Epub 2021 Dec 3. PMID 35706641
- [Background] Jensen MP, Gammaitoni AR, Olaleye DO, Oleka N, Nalamachu SR, Galer BS. The pain quality assessment scale: assessment of pain quality in carpal tunnel syndrome. J Pain. 2006 Nov;7(11):823-32. doi: 10.1016/j.jpain.2006.04.003. PMID 17074624
- [Background] Victor TW, Jensen MP, Gammaitoni AR, Gould EM, White RE, Galer BS. The dimensions of pain quality: factor analysis of the Pain Quality Assessment Scale. Clin J Pain. 2008 Jul-Aug;24(6):550-5. doi: 10.1097/AJP.0b013e31816b1058. PMID 18574365
- [Background] Hirschfeld G, Zernikow B. Variability of "optimal" cut points for mild, moderate, and severe pain: neglected problems when comparing groups. Pain. 2013 Jan;154(1):154-159. doi: 10.1016/j.pain.2012.10.008. Epub 2012 Oct 22. PMID 23182623
- [Background] Oldenmenger WH, de Raaf PJ, de Klerk C, van der Rijt CC. Cut points on 0-10 numeric rating scales for symptoms included in the Edmonton Symptom Assessment Scale in cancer patients: a systematic review. J Pain Symptom Manage. 2013 Jun;45(6):1083-93. doi: 10.1016/j.jpainsymman.2012.06.007. Epub 2012 Sep 25. PMID 23017617
- [Background] Guidelines for documentation in the gastrointestinal endoscopy setting. Society of Gastroenterology Nurses and Associates, Inc. Gastroenterol Nurs. 1999 Mar-Apr;22(2):69-97. No abstract available. PMID 10382416
- [Background] Maida M, Sferrazza S, Murino A, Lisotti A, Lazaridis N, Vitello A, Fusaroli P, de Pretis G, Sinagra E. Effectiveness and safety of underwater techniques in gastrointestinal endoscopy: a comprehensive review of the literature. Surg Endosc. 2021 Jan;35(1):37-51. doi: 10.1007/s00464-020-07907-8. Epub 2020 Aug 27. PMID 32856154